CLINICAL TRIAL: NCT05800691
Title: Predicting Factors for Mortality in Patients After the Modified Blalock-Taussig Shunt Procedure in Developing Country: a Retrospective Study
Brief Title: Predicting Factors for Mortality in Congenital Heart Disease Patients After Shunt Procedure in Developing Country.
Status: Completed | Type: Observational
Sponsor: Universitas Sumatera Utara (Other)
Collaborators: Indonesia University (Other)
Responsible Party: Principal Investigator, Putri Amelia, dr. Putri Amelia, M.Ked (Ped), Sp.A(K), Universitas Sumatera Utara
Other Study IDs: 000
Record Dates: First submitted 2023-03-12; First posted 2023-04-05 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Cyanotic Congenital Heart Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Blalock Taussig (BT) is a palliative procedure that preserves blood circulation to the lungs and alleviates cyanosis in patients with congenital heart diseases and reduced pulmonary blood flow. BT shunt remains a routinely performed procedure in developing countries before definitive surgery. However, evidence on predictors factors of mortality after this procedure is still scarce in Indonesia.

ELIGIBILITY:
Inclusion Criteria:

* All CHD pediatric patients with a previous history of BT shunt procedure.

Exclusion Criteria:

* Pediatric patients with incomplete medical records

Ages: 1 Day to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The population of this study is CHD pediatric patients with a previous history of BT shunt procedure
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
In-Hospital Mortality | November 2020 - January 2021
  Death occured to patients during in hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Sumatera Utara, Medan, North Sumatera, Indonesia